CLINICAL TRIAL: NCT02414594
Title: A Blinded, Placebo-Controlled, Dose-Escalation, Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of ISIS 681257 Administered Subcutaneously to Healthy Volunteers With Elevated Lipoprotein(a)
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IONIS APO(a)-LRx in Healthy Volunteers With Elevated Lipoprotein(a)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Collaborators: Akcea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: IONIS-APO(a)-LRx
Record Dates: First submitted 2015-04-01; First posted 2015-04-13 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Elevated Lipoprotein(a)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IONIS-APO(a)-LRx (Experimental): Drug: IONIS-APO(a)-LRx
  Interventions: Drug: IONIS-APO(a)-LRx
- Placebo (Normal Saline) (Placebo Comparator): Drug: Sterile Normal Saline (0.9% NaCl)
  Interventions: Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: IONIS-APO(a)-LRx — Ascending single and multiple doses of IONIS-APO(a)-LRx by subcutaneous (SC) injection
  Arms: IONIS-APO(a)-LRx
Drug: Sterile Normal Saline (0.9% NaCl) — Calculated volume to match active comparator
  Arms: Placebo (Normal Saline)

SUMMARY:
The purpose is to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of IONIS APO(a)-LRx (ISIS 681257) given to healthy volunteer subjects.

ELIGIBILITY:
Inclusion Criteria:

* Must have given written informed consent and be able to comply with all study requirements
* Healthy males or females aged 18-65 inclusive and weighing ≥ 50 kg at the time of informed consent
* Females must be non-pregnant and non-lactating, and either surgically sterile or post- menopausal
* Males must be surgically sterile, abstinent or using an acceptable contraceptive method
* BMI < 35.0 kg/m2
* Subjects must have Lp(a) ≥ 75 nanomoles/liter nmol/L (30 mg/dL) at Screening

Exclusion Criteria:

* Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
* Treatment with another Study Drug, biological agent, or device within one-month of screening
* Regular use of alcohol within 6 months of Screening
* Use of concomitant drugs unless authorized by the Sponsor Medical Monitor
* Smoking > 10 cigarettes a day
* Considered unsuitable for inclusion by the Principal Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single and multiple doses of IONIS-APO(a)-LRx (incidence, severity, and dose-relationship of adverse effects and changes in the laboratory parameters) | Up to 113 days
  The safety and tolerability of IONIS-APO(a)-LRx will be assessed by determining the incidence, severity, and dose-relationship of adverse effects and changes in the laboratory parameters by dose. Safety results in subjects dosed with IONIS-APO(a)-LRx will be compared with those from subjects dosed with placebo.
To evaluate the pharmacokinetics of single and multiple doses of IONIS-APO(a)-LRx (unconjugated and conjugated ASO) | Up to 113 days
  The plasma pharmacokinetics of IONIS-APO(a)-LRx (unconjugated and conjugated ASO) will be assessed following single and multiple-dose SC administration. The amount of ISIS-APO(a)-LRx excreted in urine at selected 24-hour intervals will also be determined.
To evaluate the plasma pharmacodynamics of IONIS-APO(a)-LRx (Changes in plasma Lp(a) levels) | Up to 113 days
  Changes in plasma Lp(a) levels compared to baseline.

SECONDARY OUTCOMES:
Exploratory pharmacodynamic effects of IONIS-APO(a)-LRx | Up to 113 days
  Effects of IONIS-APO(a)-LRx on changes in levels of oxidized phospholipids associated with apoB-100 compared to baseline.
Exploratory pharmacodynamic effects of IONIS-APO(a)-LRx | Up to 113 days
  Effects of IONIS-APO(a)-LRx on changes in levels of oxidized phospholipids associated with apo(a) compared to baseline.
Exploratory pharmacodynamic effects of IONIS-APO(a)-LRx | Up to 113 days
  Effects of IONIS-APO(a)-LRx on changes in Lp-PLA2 compared to baseline.
Exploratory pharmacodynamic effects of IONIS-APO(a)-LRx | Up to 113 days
  Effects of IONIS-APO(a)-LRx on changes in sPLA2 compared to baseline.
Exploratory pharmacodynamic effects of IONIS-APO(a)-LRx | Up to 113 days
  Effects of IONIS-APO(a)-LRx on changes in apo(a) isoform size compared to baseline.
Exploratory pharmacodynamic effects of IONIS-APO(a)-LRx | Up to 113 days
  Effects of ISIS-APO(a)-LRx on changes in lipid panel compared to baseline.
Exploratory pharmacodynamic effects of IONIS-APO(a)-LRx | Up to 113 days
  Effects of IONIS-APO(a)-LRx on changes in systemic markers of inflammation compared to baseline.
Exploratory pharmacodynamic effects of IONIS-APO(a)-LRx | Up to 113 days
  Effects of IONIS-APO(a)-LRx on changes in plasminogen/coagulation compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Site, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Milosavljevic MN, Stefanovic SM, Pejcic AV. Potential Novel RNA-Targeting Agents for Effective Lipoprotein(a) Lowering: A Systematic Assessment of the Evidence From Completed and Ongoing Developmental Clinical Trials. J Cardiovasc Pharmacol. 2023 Jul 1;82(1):1-12. doi: 10.1097/FJC.0000000000001429. PMID 37070852
- [Derived] Viney NJ, van Capelleveen JC, Geary RS, Xia S, Tami JA, Yu RZ, Marcovina SM, Hughes SG, Graham MJ, Crooke RM, Crooke ST, Witztum JL, Stroes ES, Tsimikas S. Antisense oligonucleotides targeting apolipoprotein(a) in people with raised lipoprotein(a): two randomised, double-blind, placebo-controlled, dose-ranging trials. Lancet. 2016 Nov 5;388(10057):2239-2253. doi: 10.1016/S0140-6736(16)31009-1. Epub 2016 Sep 21. PMID 27665230